CLINICAL TRIAL: NCT01388842
Title: Evaluation of the Efficacy and Safety of Inhaled Nitric Oxide (iNO) as Adjunctive Treatment for Cerebral Malaria in Children: A Randomized Open Label Phase II Clinical Trial
Brief Title: Evaluation of the Efficacy and Safety of Inhaled Nitric Oxide as Adjunctive Treatment for Cerebral Malaria in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Epicentre (Other)
Collaborators: Mbarara University of Science and Technology (Other); Massachusetts General Hospital (Other); Harvard Medical School (HMS and HSDM) (Other); Medecins Sans Frontieres, Netherlands (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Epicentre/MBA/2011/NO
Record Dates: First submitted 2010-11-23; First posted 2011-07-07 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-02

CONDITIONS: Malaria, Cerebral
Keywords: severe malaria; children; adjunctive treatment
MeSH Terms: conditions — Malaria, Cerebral; Malaria | interventions — Endothelium-Dependent Relaxing Factors; Nitric Oxide; Nitrogen; Air

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Controls will receive small pulses of placebo study drug via the INOpulse delivery system. Oxygen saturation will be maintained above 94% by adding oxygen to inspired gas via a loose fitting mask when necessary.
  Interventions: Drug: Placebo
- inhaled nitric oxide (Experimental): Subjects randomized to the intervention arm will receive a dose equivalent to 80 ppm iNO in air using an INOpulse delivery system for 24 hours per day for a minimum of two days and until clinical improvement (coma recovery), death or a maximum of 5 days. Oxygen saturation will be maintained above 94% by adding oxygen to inspired gas via a loose fitting mask when necessary.
  Interventions: Drug: inhaled nitric oxide

INTERVENTIONS:
Drug: inhaled nitric oxide — Study drug will be administered using an INOpulse delivery system that delivers small pulses of study drug to the patient via a nasal cannula. Subjects randomized to the intervention arm will receive a dose equivalent to 80 ppm iNO in air for 24 hours per day for a minimum of two days and until clinical improvement (coma recovery), death or a maximum of 5 days.
  Other Names: INOmax (nitric oxide) for inhalation
  Arms: inhaled nitric oxide
Drug: Placebo — The placebo will be administered using an INOpulse delivery system that delivers small pulses of study drug to the patient via a nasal cannula. Subjects randomized to the placebo arm will receive nitrogen in air for 24 hours per day for a minimum of two days and until clinical improvement (coma recovery), death or a maximum of 5 days.
  Other Names: Nitrogen in air
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess if adding inhaled Nitric Oxide to other malaria treatments can improve the outcome of cerebral malaria in children aged 2months to 12 years.

DETAILED DESCRIPTION:
Despite very effective antimalarial treatment, there is a residual and unacceptable high mortality rate of malaria, especially amongst young children. Recent progress has been made in understanding the role of Nitric Oxide (NO) in severe malaria, indicating that NO supplementation is likely to have a beneficial action in severe malaria possibly through down-regulation of inflammatory cytokines like TNF. Of the various ways to supplement NO, iNO appears to be the safest since it is very well studied in critically ill patients and does not cause systemic vasodilation. The safety of NO inhalation has been clearly demonstrated through its wide use in the treatment of persistent pulmonary hypertension in neonates and pulmonary hypertension in children and adults. Extensive data on its safety has been collected. This study is a phase 2 clinical trial that aims at demonstrating the efficacy of iNO when added to antimalarial treatment to treat cerebral malaria. This study will also provide a better understanding of the pathophysiological mechanisms involved in severe malaria.

ELIGIBILITY:
Inclusion Criteria:

* Age between 2 months and 12 years.
* With malaria infection confirmed by a malaria antigen test and/or a positive blood smear examination
* AND sustained coma: achieving a Blantyre Coma Score less than 3 for 2, or more, hours after ruling out and treating hypoglycemia (blood glucose less than 2.2 mmol/l), ruling out meningitis, and ruling out and treating active clinical seizures.

Exclusion Criteria:

* Refusal to participate
* Other cause of coma (toxic or pre-existing severe neurological disease)
* Terminal respiratory failure (due to brainstem coning)
* Coagulopathic
* Clinically unstable enough to preclude venipuncture and phlebotomy
* Severe malnutrition defined by edema or a weight-for-height minus 3 SD;
* Evidence of pre-existing brain injury
* Advanced AIDS defined by WHO clinical staging 4;

Ages: 2 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 92 (Actual)
Dates: Start 2011-09; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Angiopoietin 1 (Ang-1) | 48 hours
  Increase in Ang-1 between inclusion and 48 hours of combined therapy (iNO or placebo plus antimalarial chemotherapy)

SECONDARY OUTCOMES:
Mortality | 48 hours
  Reduction in mortality at 48 hours
coma score | 48 hours
  normalisation of coma score (Blantyre coma scale)
retinopathy | every 6 hours
  Normalisation of malaria retinopathy measured by indirect fundoscopy
tone | 48 hours
  Improvement of posture and tone
Measure of occurrence of neurological sequelae in children | months 1, 3 and 6
  Reduction of incidence of neurological sequelae, including motor dysfunction, behavioral disorders, hearing, speech and sight disorders and seizure disorders.
Vital signs | every 6 hours
  Improvement of vital signs: Systolic and diastolic blood pressure, pulse rate, temperature
oxygen saturation | every 6 hours
  Both Hb Oxygen saturation (SpO2) and total MetHb levels continuously measured by pulse oximetry (Rascal Model 7, Massimo Corp.)

CONTACTS AND LOCATIONS:
Overall Officials: Juliet Mwanga-Amumpaire, Dr, Principal Investigator — Epicentre
Locations (1):
- Mbarara Regional Referral Hospital, Mbarara, Uganda

IPD SHARING:
Plan to Share IPD: No